CLINICAL TRIAL: NCT03104322
Title: A Randomised, Crossover Study of Self-monitoring of Symptoms and Spirometry Via the patientMpower Platform in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: Patient-reported Monitoring of Symptoms and Spirometry Via the patientMpower Platform in Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: patientMpower Ltd. (Industry)
Collaborators: Health Service Executive, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IPF patientMpower 02
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Results first posted 2019-01-23 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: digital health; home spirometry; patient reported outcome measure; e-health; pirfenidone; nintedanib; FVC; antifibrotic
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Fixed-order, two-period crossover (2 x 8 weeks), no washout, usual care controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Observation sequence (Other): Period 1: patientMpower platform+usual care for 8 weeks; Period 2: usual care alone for 8 weeks
  Interventions: Other: patientMpower platform; Other: usual care

INTERVENTIONS:
Other: patientMpower platform — electronic health journal for patient to record compliance, spirometry, impact on daily life and symptoms
Other: usual care — usual care

SUMMARY:
Pilot-scale, open-label, fixed-order, two-period crossover study in idiopathic pulmonary fibrosis (IPF) over 16 weeks. Patients will use an electronic health journal (patientMpower platform) to record treatment compliance, forced vital capacity (FVC; daily), impact of IPF on daily life (weekly) and other symptoms. Objectives are to characterise acceptability of patientMpower platform from patient & healthcare professional perspective, impact of active engagement and self-monitoring using patientMpower platform on Patient Reported Outcome Measures (PROMs) in IPF, impact of patientMpower platform on medication compliance and correlation between patient-reported PROMs & FVC and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of idiopathic pulmonary fibrosis (IPF).
* daily unrestricted access to smartphone or tablet device at home.
* demonstrated understanding of protocol and correct use of Spirobank Smart spirometer and patientMpower platform.
* able and willing to perform spirometry every day at home.
* willing to give written informed consent

Exclusion Criteria:

* significant confusion or any concomitant medical condition which would limit the ability of the patient to record symptoms or use a home spirometer on a regular basis.
* new prescription of antifibrotic therapy for IPF (e.g. pirfenidone, nintedanib) within 4 weeks before baseline visit.
* recent exacerbation of IPF or other clinically significant change in the patient's medical condition in 4 weeks before baseline visit

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dept. of Respiratory Medicine, Principal Investigator — Galway University Hospital
Locations (1):
- Dept. of Respiratory Medicine, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] S. Walsh, T. Cahill, C. Edwards, E. Costello, J. Walsh, A.-M. Russell, A.W. O'Regan. Patient-Reported Monitoring of Symptoms and Spirometry Via the patientMpower Platform in Idiopathic Pulmonary Fibrosis. American Journal of Respiratory and Critical Care Medicine 2018;197: A4933

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation Sequence
Started | 7
Completed | 6
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Observation Sequence
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 69 [57 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 7
Region of Enrollment [Number; unit: participants]
  Ireland | 7

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of patientMpower Platform From Patient & Healthcare Professional Perspective
Description: Questionnaire-based assessment of response to questions: [pMp = patientMpower platform]
  1. instructions for using pMp were clear
  2. pMp helped me take the correct dose medicines
  3. pMp helped me to take my medicines at the correct time
  4. pMp helped me to reach my personal exercise goal
  5. pMp helped me to walk further
  6. pMp gave me a greater sense of control
  7. useful to be able to record the impact of lung fibrosis on QoL
  8. pMp encouraged me to look at the informational videos
  9. preference for using pMp
  10. difficulty in using pMp
  11. effect of pMp on impact on daily life
  12. tiring/irritating to use pMp
  13. want to continue using pMp after study
  14. would recommend pMp to others Possible responses Q1-8, Q12: strongly agree/agree/disagree/strongly disagree Q9: yes/no preference/no Q10: very easy/easy/difficult/very difficult Q11: positive/negative/open text Q13,14: yes/no
Time Frame: single measurement at 8 weeks
Population: Patients who completed study and provided response to questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Sequence
Number analyzed (Participants) | 4
Participants
  agree instructions clear | 3
  agree helped correct dose of meds | 1
  agree helped time of meds | 1
  agree motivated re exercise | 4
  agree helped walk further | 3
  agree gave greater sense control | 3
  agree useful record impact on QoL | 3
  agree helped look at information videos | 2
  prefer using patientMpower | 3
  easy to use patientMpower | 2
  positive effect on impact on daily life | 3
  agree tiring/irritating to use patientMpower | 0
  want to continue after end study | 4
  would recommend to others | 4

2. Secondary Outcome: Medication Compliance (Days Medication Taken/Observation Period Days)
Description: Compliance recorded by patient via patientMpower platform daily
Time Frame: 8 weeks
Population: Patients did not record medication compliance during study timeframe.
Arm/Group | Observation Sequence
Number analyzed (Participants) | 0

3. Secondary Outcome: Idiopathic Pulmonary Fibrosis Patient Reported Outcome Measure (IPF-PROM)
Description: 12-item questionnaire with 4 domains (psychological experience of dyspnoea, physical experience of dyspnoea, emotional well-being, energy levels). 3 questions/domain asking frequency of symptom or its impact in the time interval since last response. Four possible responses to each question: none of the time/some of the time/most of the time/all of the time. Numerical score assigned to each response 1/2/3/4 (respectively). Impact on domain characterised by mean score for each of 3 questions in that domain. One question on overall quality of life with responses: excellent/good/fair/poor/very poor. Numerical score assigned to each response 1/2/3/4/5 respectively. Low score better outcome; high score worse outcome (for all responses).
Time Frame: Baseline visit
Population: patients who provided at least 1 IPF-PROM; insufficient data for analysis of time trends; Baseline values reported
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Observation Sequence
Number analyzed (Participants) | 2
score on a scale
  Baseline overall quality of life | 1.5 [1 to 2]
  Baseline psychological impact of dyspnoea | 2.0 [1.3 to 2.7]
  Baseline physical impact of breathlessness | 1.85 [1.0 to 2.7]
  Baseline psychological wellbeing | 1.35 [1.0 to 1.7]
  Baseline energy | 2.0 [1.0 to 2.0]

4. Secondary Outcome: Patient-reported Exercise Performance
Description: Activity (steps/day) recorded via FitBit or patient's phone and transmitted to patientMpower platform
Time Frame: 8 weeks
Population: No data available for analysis due to technical issues (no patient used a FitBit or mobile device with built-in accelerometer)
Arm/Group | Observation Sequence
Number analyzed (Participants) | 0

5. Secondary Outcome: Patient-reported Forced Vital Capacity (FVC)
Description: Forced vital capacity recorded via patientMpower platform daily
Time Frame: 8 weeks
Population: All entered patients who provided home spirometry data
Measure: Mean (Full Range); unit: L
Arm/Group | Observation Sequence
Number analyzed (Participants) | 7
L
  Baseline FVC (patient-reported) | 2.40 [1.51 to 3.54]
  8-week FVC (patient-reported): number analyzed (Participants) | 6
  8-week FVC (patient-reported) | 2.7 [2.2 to 3.8]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Observation Sequence
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT03104322/Prot_SAP_000.pdf